CLINICAL TRIAL: NCT06159972
Title: Can EndoFLIP Improve Quality of Life Before and After Fundoplication?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Wiley Chung (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor-Investigator, Dr. Wiley Chung, Thoracic Surgeon and Assistant Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6035362
Record Dates: First submitted 2023-11-23; First posted 2023-12-07 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: GERD; Hiatal Hernia
MeSH Terms: conditions — Gastroesophageal Reflux; Hernia, Hiatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EndoFLIP (Experimental): Intraop EndoFLIP measurements
  Interventions: Device: EndoFLIP

INTERVENTIONS:
Device: EndoFLIP — EndoFLIP is a small balloon catheter that is inserted through the endoscope at the time of endoscopy.

SUMMARY:
Patients with reflux disease (heart burn), or a hiatal hernia, who do not get better with medication, may have surgery to help with their symptoms. Unfortunately, there is no agreed upon way to perform the surgery. The investigators are using a new surgical instrument called the EndoFLIP which allows surgeons to take measurements during the operation. The investigators will compare the measurements obtained during surgery with a quality of life score that we will calculate from a questionnaire.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) has a prevalence of 30% in North America (Richter 2018), where patients can present with reflux, heartburn, dysphagia, chest pain, or a combination of symptoms. Those referred by their primary care physician to a specialist have often already failed a trial of proton pump inhibitors (PPI), thus warranting further investigation. Practice guidelines from the American College of Gastroenterologists (Katz 2013) recommend that patients undergo upper endoscopy, followed by esophageal manometry, and reflux monitoring before any surgical intervention.

While these recommendations are well-founded, patient compliance with these tests remains low, since esophageal manometry and 24-hour pH testing are generally poorly tolerated, involving the placement of probes inserted nasogastrically. A qualitative study investigated patient perceptions of 24-hour pH monitoring and manometry testing (Walamies 2002) and asked 92 patients to describe their experience with manometry. Of the 84 respondents, 52% reported moderate-severe discomfort. It was shown that many patients are fearful and anxious about these tests. Some may refuse them due to their invasiveness, especially if having already undergone endoscopic evaluation. Undergoing surgery with an indeterminate diagnosis or in the absence of a full motility assessment is contraindicated by current practice guidelines and devastating consequences could occur. The lack of preoperative investigations could omit a large subset of potential surgical candidates or even lead to anti-reflux surgery in patients for the wrong diagnosis.

Once a patient is considered a surgical candidate, operative management aims to reestablish the anti-reflux barrier by plicating the gastric fundus around the gastroesophageal junction (GEJ), called fundoplication. Until now, there is no established objective measure to determine how tight to make the fundoplication. Some surgeons use a bougie to estimate the diameter of the GEJ (Patterson 2000), while some use an endoscope, and others rely on their subjective judgement. A fundoplication that is too narrow can cause severe postoperative dysphagia symptoms, whereas one that is too loose may cause recurrence or worsening of GERD symptoms. A balance is required.

The EndoFLIP balloon catheter allows users to measure the cross-sectional area (CSA), diameter, pressure and distensibility index (DI) of the GEJ. This can be done intraoperatively to obtain objective measures of the tightness of the fundoplication. These results may then be correlated with post-operative symptoms to determine the optimal CSA and DI in fundoplication. Previous studies have sought to address this problem but were limited by their lack of standardized EndoFLIP use (Su 2019). Symptom severity measurements were also captured too early in the post-operative period before a new baseline was established (Nwokedi 2020). This proposed study will have a defined EndoFLIP protocol that will be used to obtain all measurements. In addition, our post-operative readings will be captured no earlier than four months from the date of surgery. The investigators attempt to establish objective measurements to guide future operative interventions, thereby improving postoperative symptoms and overall patient satisfaction.

During the pre-operative workup, most patients with a clinical indication for 24-hour pH monitoring and manometry testing will undergo an esophagogastroduodenoscopy (EGD). This is much better tolerated, allowing for the administration of topical anesthetic and intravenous sedating medications. EndoFLIP readings can be taken at the time of EGD, thereby decreasing the number of investigations that may prolong preoperative workup. Clinicians may be able to rely on these readings alone in select patients.

Prior studies investigating the use of this novel technique have compared preoperative and post-operative CSA and DI values following a wide range of esophagogastric procedures [Attaar 2021, Ichkhanian 2020] and others have established a relationship with patient reported outcomes [Su 2020, Nwokedi 2020]. Some have compared CSA and DI in patients with and without achalasia [Carlson 2015]. Others have attempted to identify a correlation between EndoFLIP readings and anorectal manometry [Zifan 2018, Leroi 2018], and with pyloric manometry [Snape 2016]. One group of investigators [Tucker 2013] attempted to validate EndoFLIP readings with acid exposure time on pH testing and found no correlation between the two. That study was limited by its small sample size and the retrospective nature of the data, resulting in uncontrolled confounding. A true correlation between EndoFLIP measurements with 24-hour pH monitoring and esophageal manometry has yet to be identified.

To summarise, a knowledge of the intra-operative EndoFLIP measurements that correlate with acceptable post-operative symptom severity scores will be useful information for surgeons performing a fundoplication (there currently is no gold standard for fundoplication creation). Secondly, if pre-operative EndoFLIP measurements correlate well with pre-operative 24-hr pH studies and manometry testing, then there is a potential for EndoFLIP to replace these invasive, uncomfortable, and poorly tolerated tests. This may result in increased patient compliance and reduced costs of pre-operative testing.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing workup for gastroesophageal reflux disease (GERD) and/or symptomatic hiatal hernia who undergo fundoplication AND who undergo fundoplication

Exclusion Criteria:

* Those with a previous history of hiatal hernia repair, fundoplication, esophagectomy, or gastrectomy
* Inability to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-05 (Actual); Primary Completion 2024-07-05 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Intraoperative EndoFLIP and postoperative quality of life using the "GERD health related quality of life" score | 4 (four) months
  To identify the correlation between intra-operative EndoFLIP measurements of cross-sectional area, distensibility index, and contraction pattern with post-operative symptom severity score for GERD using the "GERD health related quality of life" score.

SECONDARY OUTCOMES:
Intraop EndoFLIP and preop + postop manometry and pH monitoring | 4 (four) months
  To identify the correlation between intra-operative EndoFLIP measurements of cross-sectional area, distensibility index with 24-hour pH monitoring, before and after fundoplication; and to identify a correlation between contraction pattern and manometry before and after fundoplication.

CONTACTS AND LOCATIONS:
Overall Officials: Wiley Chung, MD MHPE, Principal Investigator — Queen's University
Locations (1):
- KHSC, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No